CLINICAL TRIAL: NCT04770909
Title: Log2Lose: Incenting Weight Loss and Dietary Self-monitoring in Real-time to Improve Weight Management Among Adults With Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Duke University (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 2020-1693; A539722 (Other: UW Madison); SMPH/SURGERY (Other: UW Madison); Protocol Version 1/3/2025 (Other: UW Madison); UG3HL150558-01 (NIH)
Record Dates: First submitted 2021-02-22; First posted 2021-02-25 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: 2 (incentives for dietary self-monitoring: yes vs. no) x 2 (incentives for weight loss: yes vs. no)
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Combined (Experimental): Weekly incentives for dietary self-monitoring and weight loss
  Interventions: Behavioral: Incentives for dietary self-monitoring and weight loss
- Dietary self-monitoring (Experimental): Weekly incentives for dietary self-monitoring
  Interventions: Behavioral: Incentives for dietary self-monitoring
- Weight loss (Experimental): Weekly incentives for weight loss
  Interventions: Behavioral: Incentives for weight loss
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Incentives for dietary self-monitoring and weight loss — Participants can earn up to $300 during the trial for achieving adequate dietary self-monitoring and weight loss
  Arms: Combined
Behavioral: Incentives for dietary self-monitoring — Participants can earn up to $300 during the trial for achieving adequate dietary self-monitoring
  Arms: Dietary self-monitoring
Behavioral: Incentives for weight loss — Participants can earn up to $300 during the trial for achieving weight loss
  Arms: Weight loss

SUMMARY:
This study involves an evaluation of whether providing small incentives weekly for dietary self-monitoring and/or weight loss improves short- and long-term weight loss. Participants can expect to be on study for 18 months.

DETAILED DESCRIPTION:
In this two-site, randomized, single-masked, longitudinal 2x2 factorial study, called Log2Lose, adults with obesity from Madison, WI and Durham, NC will be offered a 78 week, evidence-based behavioral weight management program comprising an incentivized weight loss intervention for 26 weeks (Phase I), an incentivized weight loss maintenance intervention for 26 weeks (Phase II), and a non-incentivized weight maintenance intervention for 26 weeks (Phase III). Participants will be randomized in a 2x2 design to receive adjunctive incentives for either weekly weight loss or dietary self-monitoring, both, or neither. The investigators will assess the proportion of participants achieving clinically significant weight loss of greater than or equal to 5 percent at the end of each phase.

All participants will participate in an 18-month weight management program delivered via videoconference.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥30 kg/m2
* Desire to lose weight
* Agrees to attend outcome visits per protocol
* Available for class times
* Transportation and ability to attend in-person study visits at baseline (screening), 26, 52, and 78 weeks
* Able to stand for weight measurements without assistance
* Able to speak and read English
* Able to download and use the MyFitnessPal and Fitbit apps daily
* Possess smart phone with data and texting plan
* Have or willing to create a Gmail address
* Able to connect to a video conference call using a smartphone, tablet or computer with a webcam and microphone
* Score of at least 4 out of 6 on a validated cognitive screener

Exclusion Criteria:

* Weight >380 lb
* Weight loss of at least 10 lbs in the month prior to screening
* Currently enrolled or enrolled in previous month in a clinical, research, or community program focusing on lifestyle change that could affect weight
* Current use of weight loss medication
* History of bariatric surgery or planning to have bariatric surgery in the study timeframe
* Residing in a nursing home or receiving home health care
* Impaired hearing
* Significant dementia, drug or alcohol misuse, or unstable psychiatric illness (e.g., schizophrenia, psychosis)
* Current treatment for cancer or being treated for cancer (besides basal cell carcinoma or squamous cell) in the last 6 months
* Use of insulin, sulfonylureas, or meglitinides due to increased risk for hypoglycemia
* Pregnant, breastfeeding, or planning to become pregnant within the study timeframe
* Diuretic medication doses higher than hydrochlorothiazide 25 mg daily, furosemide 40 mg daily, torsemide 20 mg daily, bumetanide 1 mg daily, or any use of metolazone; use of potassium-sparing diuretics is acceptable
* Chronic kidney disease at stage 4 or 5
* Unstable heart disease in the 6 months prior to screening
* Exertional chest pain
* History of ascites requiring paracentesis
* Pain, fainting or other conditions that prohibit mild/moderate exercise

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 706 (Actual)
Dates: Start 2021-05-13 (Actual); Primary Completion 2024-04-08 (Actual); Study Completion 2025-04-10 (Actual)

PRIMARY OUTCOMES:
Percent of participants who achieve clinically significant weight loss of at least 5 percent of baseline weight at 26 weeks | 26 weeks
  Measured on a calibrated, digital scale to the nearest 0.1 kg

SECONDARY OUTCOMES:
Percent of participants who achieve clinically significant weight loss of at least 5 percent of baseline weight at 52 weeks | 52 weeks
  Measured on a calibrated, digital scale to the nearest 0.1 kg
Percent of participants who achieve clinically significant weight loss of at least 5 percent of baseline weight at 78 weeks | 78 weeks
  Measured on a calibrated, digital scale to the nearest 0.1 kg
Change in dose equivalents of cardiovascular medications from baseline to 78 weeks | Baseline, 78 weeks
  Dose equivalents for antihypertensive, antilipemic, and type 2 diabetes medications
Change in diastolic blood pressure from baseline to 26, 52, and 78 weeks | Baseline, 26, 52, and 78 weeks
  Average of two sequential measurements measured on a digital blood pressure monitor. A second reading will be taken one minute after the first. If the difference between the systolic measurements is greater than 15mmHg, then a third reading will be taken, one minute after the second reading.
Change in systolic blood pressure from baseline to 26, 52, and 78 weeks | Baseline, 26, 52, and 78 weeks
  Average of two sequential measurements measured on a digital blood pressure monitor. A second reading will be taken one minute after the first. If the difference between the systolic measurements is greater than 15mmHg, then a third reading will be taken, one minute after the second reading.

OTHER OUTCOMES:
Intrinsic motivation for weight loss as assessed by modified Treatment Self-Regulation Questionnaire | 26 weeks
  Association of intrinsic motivation for weight loss with proportion of patients who achieve clinically significant weight loss of at least 5 percent of baseline weight at 26 weeks will be measured with modified version of Treatment Self-Regulation Questionnaire. Intrinsic motivation will be calculated as mean of items 2, 4, 6, 8, 11, 14, 16, 17. Each item can be answered from '1 - not at all true' to '6 - very true'. Lower scores correspond to lower intrinsic motivation for weight loss
Extrinsic motivation for weight loss as assessed by modified Treatment Self-Regulation Questionnaire | 26 weeks
  Association of extrinsic motivation for weight loss with proportion of patients who achieve clinically significant weight loss of at least 5 percent of baseline weight at 26 weeks will be measured with modified version of Treatment Self-Regulation Questionnaire.
  Extrinsic motivation will be calculated as mean of items 1, 3, 5, 7, 9, 10, 12, 13, 15, 18. Each item can be answered from '1 - not at all true' to '6 - very true'. Lower scores correspond to lower extrinsic motivation for weight loss

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Cadmus-Bertram, PhD, Principal Investigator — University of Wisconsin, Madison; Corrine Voils, PhD, Principal Investigator — University of Utah Department of Internal Medicine
Locations (2):
- United States (2):
  - Duke University Medical Center, Durham, North Carolina
  - University of Wisconsin-Madison, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
First, investigators will strip all data of personal identifiers (i.e., personal health information (PHI)) in accordance with the HIPAA privacy rule. Each consented and enrolled participant will be assigned a unique study ID, which will be the only participant-level identifier. Time information starting at baseline will be coded in units of study time, with baseline = '0' and termination of 18 months or dropout for all participants, regardless of the calendar date of their baseline visit. Proprietary software code will be shared in accordance with institutional policies and consent of the creators.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Study data will be made available for use by investigators not associated with the proposed study within three years after the primary results have been published.
Access Criteria: 1. The data will be used for research or implementation purposes and not to identify individual participants
  2. The data must be secured using the appropriate computer technology
  3. The data must be destroyed or returned after analyses are complete
  4. The authors of any manuscript resulting from the Log2Lose data must acknowledge the source of the data upon which their manuscript is based.
  5. Any analyses for the purpose of presentation, abstracts, and/or publications must be coordinated with the Log2Lose leadership team, so there can be some coordination of analyses to ensure that redundant analyses are not being performed independently
  6. All coauthors must be given an opportunity for review and approval of a draft manuscript prior to submission for publication.

REFERENCES:
- [Derived] Shaw RJ, Miller H, Barnes C, Davenport C, Morton-Oswald S, Jackson S, Bean M, Cohen J, Griffin C, Pendergast J, Olsen M, Gierisch J, Voils C. Development, Challenges, and Evolution of the Log2Lose Intervention for Weight Management: Randomized Controlled Digital Health Trial. JMIR Form Res. 2025 Nov 17;9:e70842. doi: 10.2196/70842. PMID 41248493
- [Derived] Voils CI, Gierisch JM, Pendergast JF, Davenport CA, Olsen MK, Barnes C, Bean M, Cadmus-Bertram L, Colon J, Elwert F, Garza K, Gavin KL, Jackson S, Miller H, Morton-Oswald S, Pabich S, Reed SD, Yancy WS Jr, Shaw RJ. Study protocol for Log2Lose: A randomized controlled trial to evaluate financial incentives for dietary self-monitoring and interim weight loss in adults with obesity. Contemp Clin Trials. 2025 Sep;156:108042. doi: 10.1016/j.cct.2025.108042. Epub 2025 Aug 5. PMID 40774423

DOCUMENTS (1):
  • Informed Consent Form (2023-08-08): https://cdn.clinicaltrials.gov/large-docs/09/NCT04770909/ICF_001.pdf